CLINICAL TRIAL: NCT01249326
Title: Protein Need and Interest of " Quick Proteins " to the Obese Subject Operated by Bariatric Surgery (BIBOP)
Acronym: BIBOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Hospices Civils de Lyon (Other); Service de médecine du Sport et des Explorations Fonctionnelles - CHRU de Clermont-Ferrand (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-0084; 2009-A01093-54 (Registry Identifier: Afssaps)
Record Dates: First submitted 2010-11-15; First posted 2010-11-29 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Morbid obesity,; Bariatric surgery, by-pass, sleeve gastrectomy,; Nitrogen balance,; Protein requirement,; Weight loss; Muscle wasting, muscle disability
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss; Muscular Atrophy | interventions — Bariatric Surgery

INTERVENTIONS:
Other: bariatric surgery — This is a prospective longitudinal study of the effect of bariatric surgery on protein requirements and protein metabolism, and protein supplementation interest, appropriate to the digestive tract changes, for the mass and muscle function

SUMMARY:
The main objective of the study is to evaluate the protein requirement associated with postoperative weight loss caused by by-pass (shunt which leads to a certain degree of malabsorption) or sleeve gastrectomy (more technically conservative with less malabsorption), through the study of nitrogen balance. The benefit of protein supply easily absorbed and with high essential amino acids content (proteins "fast" soluble milk) on protein metabolism and muscle function will also be studied. Endotoxemia and intestinal flora variations were measured before and after bariatric surgery.

DETAILED DESCRIPTION:
This is a prospective longitudinal study of the effect of bariatric surgery on protein requirements and protein metabolism, and protein supplementation interest, appropriate to the digestive tract changes, for the mass and muscle function. Three groups of patients will be studied: One group undergoing sleeve gastrectomy in Clermont-Ferrand (group 1: n = 20) will be followed by current recommendations. A second group undergoing sleeve gastrectomy in Clermont-Ferrand (group 2: n = 20) will receive during three months, protein supplement (powder whey protein ("fast")) at dose of 40g / day. 10 patients in group 1 and 10 patients in group 2 will participate in protein metabolism study. The third group undergoing gastric bypass in Lyon (group 3: n = 20) will be followed by the current recommendations and will participate in study of endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

- Males and females.

* Age between 18 to 60 years.
* Body mass index: BMI> 40 kg/m2,
* Biological Review considered satisfactory by the investigator based on the topics covered
* Serology HIV ( Human Immunodeficiency Virus )and HCV (Hepatitis C Virus ) negative.
* Subject giving his written informed consent
* Affiliated to National Health Insurance

Exclusion Criteria:

* Subject under 18 or over 60 years.
* Balance Organic considered abnormal by the investigator.
* Serology HIV or HCV positive.
* Pregnant or lactating.
* For women of childbearing age: β-HCG assay positive and not having reliable contraceptives (oral contraceptive, IUD (Intrauterine Device), implant or hormone patch, abstinence).
* Medical or surgical history (judged by investigator to be incompatible with the study).
* Subject with unstable psychiatric condition
* Blood donation in the two months preceding the study.
* Heavy alcohol consumption (> 2 to 3 glasses per day depending on sex) or presence of an addiction.
* Tobacco significant (> 5 cigarettes / day or equivalent in cigars or pipe tobacco).
* Subjects with an allergy or intolerance to dairy products.
* Intense sporting activity (> 5 hours / week).
* Being in exclusion on the National Volonteers Data file or having perceived more than 4500 Euros in the year for clinical study participation.
* No one under guardianship or not subject to social security.
* Subjects deprived of their liberty by judicial or administrative decision.
* Refusal to sign the information sheet and written consent for participation
* Subject with a cardiovascular or neoplasic evolutive disease
* Subject with a severe infection in the 3 months period before inclusion (assessed by doctor during inclusion consultation)
* Hypercorticism and dysthyroïdism
* Subject with a known neuro-muscular disease
* Subject with a chronic or acute inflammatory disease in the 3 months period before inclusion
* Subject treated by: corticoids, immunosupressor, anabolic agents, growth factor or having stopped treatment for less than 3 months before inclusion.

Furthermore for subjects having undergone a by-pass at Lyon:

* Subject consuming pre or probiotics many times per day, having an impact on intestinal flora.
* Subject with antibiotics during the 3 months before the beginning of the study.
* Subject with an intolerance to dairy products and refusing to consume dairy prod

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2015-03-19 (Actual)

PRIMARY OUTCOMES:
to measure the nitrogen balance and its variation during weight loss | before, after 3 months and 1 year after the operation

SECONDARY OUTCOMES:
Protein metabolism of body and muscle will be assessed | before and 3 months after surgery
- Body composition will be assessed using deuterated water (2H2O) ingested and by BIA (Bioelectrical Impedance Analysis ) | before, after 3 months and 1 year after surgery
Changes of endotoxemia will be assessed by measuring blood levels of endotoxin, their carriers, inflammatory cytokines, and protein transfer fasting and after a high fat breakfast test | before and 3 months after surgery
The voluntary muscular force and muscular weariness will be assessed in Clermont-Ferrand and Lyon by Dynatrac measurement apparatus | before, after 3 months and 1 year after the operation
Muscle mass will be estimated by urinary creatinine measurements | before, after 3 months and 1 year after the operation).
Intestinal flora microbiology analysis will be performed | 3 months and 1 year after bariatric surgery
Daily physical activity will be measured by an Acti-Heart apparatus | before, after 3 months and 1 year after surgery
- Insulino-resistance will be measured by the HOMA test( test aHomeostatic Model Assessment)and the DISSE index ((Disse E, Diabetes & Metabolism, 2008). | before, after 3 months and 1 year after surgery)
Inflammatory, hormonal, metabolic parameters' variation will be assessed by blood biological and urinary parameters measurement | before, after 3 months and 1 year after surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Guillet C, Masgrau A, Mishellany-Dutour A, Blot A, Caille A, Lyon N, Pereira B, Slim K, Robert M, Disse E, Feugier N, Le Ruyet P, Louvet C, Miolanne M, Farigon N, Laville M, Boirie Y. Bariatric surgery affects obesity-related protein requirements. Clin Nutr ESPEN. 2020 Dec;40:392-400. doi: 10.1016/j.clnesp.2020.06.007. Epub 2020 Oct 1. PMID 33183568